CLINICAL TRIAL: NCT05480748
Title: Oxygen Reserve Index in Predicting Hypoxemia in Morbidly Obese Patients
Brief Title: Oxygen Reserve Index Predicting Hypoxemia
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gülten Arslan, Assoc Dr, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: DrLutfiKirdarANEST
Record Dates: First submitted 2022-06-23; First posted 2022-07-29 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Oxygen Deficiency; Apnea
Keywords: Oxygen reserve index,; Tolerable apnea time,; Oxygen reserve index warning time,; Preoxygenation,; Percutaneous oxygen saturation warning time
MeSH Terms: conditions — Hypoxia; Apnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: 19>BMI<25 AND BMI>40: 51 patients with BMI>40 kg/m2 (morbidly obesity) and 51 patients with 19<BMI<25 kg/m2 (normal BMI), 18-75 aged, American Society of Anesthesiologists (ASA) physical status I-III scheduled for an elective surgical procedure requiring general anesthesia with endotracheal intubation.
  Interventions: Device: monitoring
- Normal body mass index and morbidly obese groups: 51 patients with BMI>40 kg/m2 (morbidly obesity) and 51 patients with 19<BMI<25 kg/m2 (normal BMI), 18-75 aged, American Society of Anesthesiologists (ASA) physical status I-III scheduled for an elective surgical procedure requiring general anesthesia with endotracheal intubation.
  Interventions: Device: monitoring

INTERVENTIONS:
Device: monitoring — ORI warning time, SpO2 warning time, added time were recorded.

SUMMARY:
After obtaining the approval of the hospital ethics committee, this prospective, observational study included written informed consent from 51 participants with 19<BMI<25 m/kg2 and 51 participants with BMI>40 m/kg2 undergoing an elective surgical requiring endotracheal intubation. In addition to standard monitors, an oxygen reserve index (ORI) sensor was placed and baseline values were recorded. The participants were preoxygenated until end expiratory oxygen concentration (EtO2) is reached 90%. After anesthesia induction and endotracheal intubation, the breathing circuit was not connected endotracheal tube until the peripheral oxygen saturation (SpO2) decreased until 95%.ORİ and SpO2 values were continuously recorded. Time of tolerable apnea, ORI warning, SpO2 warning and added warning were also recorded.

DETAILED DESCRIPTION:
This single-center prospective, observational study was approved by Institutional Ethics Committee (Decision No:2022/514/222/9, Date:30/03/2022) and was performed in accordance with the Declaration of Helsinki. Written, informed consent was obtained from 51 participants with BMI>40 kg/m2(morbidly obesity) and 51 participants with19<BMI<25 kg/m2(normal BMI), 18-75 aged, American Society of Anesthesiologists (ASA) physical status I-III scheduled for an elective surgical procedure requiring general anesthesia with endotracheal intubation. Participants with significant history of cardiopulmonary disease, 25<BMI<40 kg m2, ASA>4 and<18 years of age, difficult intubation, pregnancy, hemoglobinopathies and preoperative hemoglobin of less than 10.0 mg/dL were defined as exclusion criteria.

Standard monitors were routinely established for each participants, including heart rate (HR), noninvasive blood pressure measurements. In addition, an ORi and SpO2 were measured simultaneously at 1-s interval with a pulse oximetry sensor (Rainbow sensor, R2-25) applied to the finger and connected to a Masimo Root with Radical-7 pulse oximeter (Masimo Corp.) Data for analysis was downloaded from the Root monitor.

Following the placement of monitors, baseline values were recorded. Participants were then preoxygenated with spontaneous ventilation and 100% inspirative oxygen concentrate (FiO2) at a flow rate of 8 liter/minute via a tight-fitting face mask until EtO2 is reached to 90%. Anesthesia was induced with intravenous midazolam, fentanyl, propofol and rocuronium in 100% FiO2.The trachea was intubated after 3-4 minutes under direct visualization using a videolaryngoscope to confirm placement.The endotracheal tube was not connected to the breathing circuit, and the participants remained apneic. The World Health Organization defines intraoperative SpO2 ≥ 95% as normal in its training materials, and treatment steps are mentioned for SpO2 ≤ 94% [12]. However, since we included morbidly obese participants with limited functional residual capacities in our study and wanted to stay with in the safe range, we allowed SpO2 to decrease up to 95%. At the same time, the alarm point for SpO2 is applied as 95% in our clinic's protocol for morbidly obese patients.

ORi and SpO2 values were recorded continuously. Subsequently, the anesthesia circuit was connected and patients were ventilated with 100% Fraction of Inspired Oxygen ( FiO2), tidal volume targeted 7 ml/kg and 5 cmH2O of positive end-expiratory pressure until ORi plateaued.Thereafter, anesthesia continued per routine.

ORi and SpO2 data were compared at five specific time points: 1) baseline; 2) at the end of pre-oxygenation when the EtO2 reaches to 90%; 3) at the beginning of intubation; 4) when SpO2 reaches 95%; and 6) during ventilation with 100% FiO2 when the ORi reaches a plateau.

Investigators also recorded the tolerable apnea time defined as the time from the beginning of apnea until SpO2 reached 95% and ventilation was reinstated. The ORi warning time was defined as the time between the onset of the ORi and the SpO2 reaching 95%. Investigators defined the SpO2 warning time as the time for SpO2 to decrease from 97% to 95%.The added warning time provided by ORi was defined as the difference between ORi warning time and SpO2 warning time The time at which the ORi alarm. Alarm activation was based on the fractional rate of change in ORi rather than on a specific oxygen reserve value.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years,
* ASA 1-3,
* BMI>40 kg/m2 (morbidly obesity)
* 19<BMI<25 kg/m2 ,
* Elective surgical procedure requiring general anesthesia with endotracheal intubation

Exclusion Criteria:

* History of cardiopulmonary disease,
* 25<BMI<40 kg m2,
* <18 years of age,
* Difficult intubation,
* Pregnancy,
* Hemoglobinopathies
* Preoperative hemoglobin of less than 10.0 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 102 patients, ASA 1-3, 18-75 years
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
In morbidly obese patients oxygen reserve index (ORi) warning time, SpO2 warning time, and added warning time defined as the difference between the two to set deadlines in specific time periods. | 'Time until ORI reaches to 0.24 (It is evaluated in the first 15 minutes after the patient is given anesthesia)
  Primary endpoint; To evaluate whether ORi provides an earlier, more relevant clinical warning of impending desaturation compared to pulse oximetry in morbidly obese patients.

SECONDARY OUTCOMES:
In morbidly obese patients oxygen reserve index (ORi) warning time, SpO2 warning time, and added warning time defined as the difference between the two to set deadlines in specific time periods. | Time until SpO2 drops to 95% after ORi reaches 0.24 (until 30 minutes)
  secondary endpoint was; to compare the added warning time in patients with normal body mass index (BMI) and morbid obesity.
In morbidly obese patients oxygen reserve index (ORi) warning time, SpO2 warning time, and added warning time defined as the difference between the two to set deadlines in specific time periods. | Time from intubation until SpO2 drops to 95% (until 30 minutes)
  secondary endpoint was; to compare the tolerable apne time in patients with normal body mass index (BMI) and morbid obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Gülten Arslan, Dr, Principal Investigator — University of Health science Kartal Dr Lütfi Kırdar Training and Research Hospital
Locations (1):
- University of Health Science, Kartal Dr Lütfi Kırdar Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will share the parameters and results of the study.

REFERENCES:
- [Result] Fleming NW, Singh A, Lee L, Applegate RL 2nd. Oxygen Reserve Index: Utility as an Early Warning for Desaturation in High-Risk Surgical Patients. Anesth Analg. 2021 Mar 1;132(3):770-776. doi: 10.1213/ANE.0000000000005109. PMID 32815872
- [Result] Tsymbal E, Ayala S, Singh A, Applegate RL 2nd, Fleming NW. Study of early warning for desaturation provided by Oxygen Reserve Index in obese patients. J Clin Monit Comput. 2021 Aug;35(4):749-756. doi: 10.1007/s10877-020-00531-w. Epub 2020 May 18. PMID 32424516
- [Derived] Saracoglu KT, Arslan G, Saracoglu A, Sezen O, Ratajczyk P, Gaszynski T. Oxygen reserve index vs. peripheral oxygen saturation for the prediction of hypoxemia in morbidly obese patients: a prospective observational study. BMC Anesthesiol. 2024 Oct 11;24(1):367. doi: 10.1186/s12871-024-02755-8. PMID 39394112